CLINICAL TRIAL: NCT05956912
Title: Implementing Group Metacognitive Therapy in Cardiac Rehabilitation Services (PATHWAY-Beacons)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manchester (Other)
Collaborators: Greater Manchester Mental Health NHS Foundation Trust (Other); University of York (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Adrian Wells, Professor of Clinical and Experimental Psychopathology, University of Manchester
Other Study IDs: IRAS ID: 313677; 29567 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2023-05-09; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Anxiety; Depression; Cardiac Rehabilitation
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Cardiac rehabilitation (CR) services aim to improve heart disease patients' health and quality of life and reduce the risk of further cardiac events. Depression and anxiety are common among CR patients, and current psychological treatments for cardiac patients have minor effects. However, the NIHR-funded PATHWAY trial found that group Metacognitive Therapy (MCT) was associated with improvements in anxiety and depression when added to CR and was more effective than usual CR alone. Group MCT was also associated with preventing anxiety and depression. The next steps will establish beacon sites for delivering MCT and pilot-test additions to the national audit of cardiac rehabilitation (NACR) data capture mechanism to include an MCT data field. Such steps will support a quantitative and qualitative evaluation of implementation.

Methods: The investigators aim to address questions concerning the quality of patient data recorded, level of adoption at sites, the characteristics of patients attending MCT, the impact of adding MCT to CR on mental health outcomes, and patient, healthcare staff and commissioner views of barriers/enablers to implementation. The investigators will deliver training in group MCT to CR staff from CR services across England. The investigators will conduct semi-structured qualitative interviews with CR staff trained in group MCT to assess views on the training programme, including successes and barriers to implementation of training and delivery. The investigators will interview 8-10 CR stakeholders to identify any barriers to implementation and how these might be resolved.

Discussion: The study will support development of an NHS roll-out strategy and systematic data collection that can be used to evaluate wide-scale implementation. The study can benefit service users by improving patients' mental health outcomes and CR practitioners' clinical skills. Results will be disseminated via peer-reviewed journals, national and international conferences and service user/voluntary sector organisations and networks.

ELIGIBILITY:
Qualitative Inclusion Criteria:

All CR staff must meet the following inclusion criteria to be eligible:

1. Be a healthcare professional working with cardiac rehabilitation services being trained to deliver group-MCT
2. Be a healthcare professional working with cardiac rehabilitation or be a professional working at the commissioner level
3. Minimum of 18 years old
4. Competent level of English Language skills (able to read, understand and complete interviews in English).

Exclusion Criteria:

1. Below 18 years of age
2. Not a healthcare professional or professional working at the commissioner level
3. Does not have a competent level of English language skills

Audit inclusion criteria:

All patients attending CR who meet the NICE recommendations for acute coronary syndrome (NG185) and heart failure (NG106) will be offered group MCT as part of routine CR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cardiac rehabilitation staff trained in delivering Group-MCT, wider cardiac rehabilitation staff and managers, and healthcare professionals from local clinical commissioning groups.
  All CR patients attending cardiac rehabilitation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Adoption of group MCT | Within the 6 months that MCT is being delivered in CR services
  Successful adoption of group MCT at each site is set a-priori. A traffic-light criteria will be used to determine successful adoption.
  1. Green - achieved all of the following: a) Delivered two 6-session group MCT courses (b) at least three patients per group, and (c) a combined total of at least 60% attending four or more sessions.
  2. Amber - achieved one of the three criteria given above.
  3. Red - achieved none of the criteria.
  A Green rating indicates that a site has fully met the criteria for successful adoption. Red indicates a failure to meet the requirements. Amber is partial adoption, where amendments to procedures and protocols might lead to successful adoption. At Amber sites, specific qualitative work will be undertaken to understand the reasons for not meeting criteria more fully and to help develop strategies to ameliorate this. An overall assessment will be made considering the traffic-light ratings of all six beacon sites.

SECONDARY OUTCOMES:
Dartmouth Coop | Initial Cardiac Rehabilitation Assessment (Baseline) & Within 6 months of attending cardiac rehabilitation (Discharge)
  The COOP will be captured through the National Audit for Cardiac Rehabilitation. It is a self-report measure designed to evaluate the functional abilities of medical patients. It consists of nine items covering various areas such as physical function, daily activities, pain, social activities, social support, emotions, overall health, changes in health, and quality of life. Each chart includes text and illustrations to assist the user in responding. The responses are graded on an ordinal scale of 1 to 5, with one being the best score.
Semi-structured interviews will explore the views and opinions of group-MCT in CR (CR staff trained in group-MCT) | 1 month prior to training in MCT
  To understand what CR staff views of training in group MCT are with a view to understanding enablers and barriers. To understand the consequences, both expected and unexpected, of implementing group-MCT, for example on existing CR services, staffing needs, administration and resource requirements.
Semi-structured interviews will explore the views and opinions of group-MCT in CR (CR staff trained in group-MCT) | Within 1 month of delivering the pilot group of MCT
  To understand what CR staff views of training in group MCT are with a view to understanding enablers and barriers. To understand the consequences, both expected and unexpected, of implementing group-MCT, for example on existing CR services, staffing needs, administration and resource requirements.
Semi-structured interviews will explore the views and opinions of group-MCT in CR (CR staff trained in group-MCT) | Upon completion of delivering group-MCT, approximately 5 months after starting the delivery of MCT in CR
  To understand what CR staff views of training in group MCT are with a view to understanding enablers and barriers. To understand the consequences, both expected and unexpected, of implementing group-MCT, for example on existing CR services, staffing needs, administration and resource requirements.
Semi-structured interviews will explore the views and opinions of group-MCT in CR (CCG and other management stakeholders) | Through implementation of MCT in CR services, approximately 7 months.
  To understand the acceptability and feasibility of roll-out at commissioner level and what the enablers or barriers are. To understand the consequences, both expected and unexpected, of implementing group-MCT, for example on existing CR services, staffing needs, administration and resource requirements.
Hospital Anxiety and Depression Scale (HADS) | Initial Cardiac Rehabilitation Assessment (Baseline) & Within 6 months of attending cardiac rehabilitation (Discharge)
  The HADS will be captured through the National Audit for Cardiac Rehabilitation. It is a 14-item self-report questionnaire that measures symptoms of anxiety (7 items) and depression (7 items). Items are rated using a 4-point (0-3) scale, with higher scores indicating elevated distress. Scores for each subscale range from 0 to 21 and can be categorised as normal (0-7), mild (8-10), moderate (11-14), or severe (15-21).

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Wells, PhD, Principal Investigator — University of Manchester
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

REFERENCES:
- [Derived] Wells A, Reeves D, Belcher A, Wilson P, Doherty P, Capobianco L. Protocol for an implementation study of group metacognitive therapy for anxiety and depression in NHS cardiac rehabilitation services in England (PATHWAY-Beacons). Front Health Serv. 2024 Oct 17;4:1296596. doi: 10.3389/frhs.2024.1296596. eCollection 2024. PMID 39483442
- See also: Research Project Website Page — https://adept-ru.com/research-projects/pathway-beacons/